CLINICAL TRIAL: NCT03181672
Title: Influence of Stellate Ganglion Block on Tourniquet Response in Lower Limbs.
Brief Title: Stellate Ganglion Block on Tourniquet Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2017-KL012-01
Record Dates: First submitted 2017-06-01; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Stellate Ganglion Block
Keywords: Stellate ganglion block Tourniquet reaction
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block (Active Comparator): Stellate ganglion block
  Interventions: Procedure: Stellate ganglion block
- control group (Placebo Comparator): Deltoid muscle injection
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: Stellate ganglion block — Stellate ganglion block with 1% lidocaine 10ml
  Arms: Stellate ganglion block
Procedure: control group — Deltoid muscle injection with 1% lidocaine 10ml
  Arms: control group

SUMMARY:
To investigate the influence of stellate ganglion block on tourniquet response during surgery in patients undergoing elective lower limb Department of orthopedics.

DETAILED DESCRIPTION:
Select elective general anesthesia in 100 cases of lower extremity Department of orthopedics surgery patients were randomly divided into SGB group and control group, SGB group received anesthesia before the right stellate ganglion block intervention, the control group underwent right deltoid muscle injection, changes in hemodynamics in two groups were recorded in heart rate, blood pressure, and before anesthesia, after intubation 3min 1H, a tourniquet, tourniquet release before and after tourniquet release 3min, 30min, changes in blood physiological analysis. The effect of stellate ganglion block on tourniquet response during perioperative period was observed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anesthesiologists Grade 1-3 Patients
* undergoing lower limb surgery under general anesthesia
* should be treated with tourniquet

Exclusion Criteria:

* Tourniquet application time is less than 1h, greater than 1.5h
* Abnormal coagulation function
* perioperative application of hormone
* lidocaine allergy
* can not cope with nerve block
* nerve block failure
* minimally invasive surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 2 hours in perioperative period
  mmHg
heart rate | 2 hours in perioperative period
  bpm
Lac | One minute after the radial artery puncture, the tourniquet was applied for 1 hours and the tourniquet was released 3 minutes after the tourniquet release 30 minutes
  blood gas analysis mmol/L
cortisol | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA ng/ml
norepinephrine | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA nmol/L
(untitled outcome) | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  n nitrate reductase method μmol/L
ET-1 | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA ng/L
MDA | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA nmol/ml
SOD | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA μg/L
IL-6 | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA pg/ml
cTn-T | One minute after the radial artery puncture, one minute after intubation, tourniquet application 1 hour, one minute before tourniquet, loose after a tourniquet for 3 minutes, 30 minutes after a tourniquet
  ELISA μg/L
postoperative pain | hour 1、hour 6、hour 24、hour 48 after operation
  VAS score

SECONDARY OUTCOMES:
Complication of puncture | 2 hours in perioperative period
  bleeding、nerve injury、

CONTACTS AND LOCATIONS:
Overall Officials: Tie Xu, MD, Study Director — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published.

REFERENCES:
- [Background] Arai YC, Ogata J, Matsumoto Y, Yonemura H, Kido K, Uchida T, Ueda W. Preoperative stellate ganglion blockade prevents tourniquet-induced hypertension during general anesthesia. Acta Anaesthesiol Scand. 2004 May;48(5):613-8. doi: 10.1111/j.0001-5172.2004.00389.x. PMID 15101858